CLINICAL TRIAL: NCT00198523
Title: A Multi-Center, Randomized, Double Masked, Bioequivalence Study of Tobramycin and Prednisolone Acetate (0.3/1.0%, ISTA) Ophthalmic Suspension Compared to PredForte (1.0% Prednisolone Acetate, Allergan) Ophthalmic Suspension
Brief Title: A Bioequivalence Study of Tobramycin and Prednisolone Acetate Compared to PredForte
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-TP-CPK01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Eye Infections; Postoperative Complications
Keywords: Cataract Extraction; Anti-Bacterial Agents; Steroids
MeSH Terms: conditions — Eye Infections; Postoperative Complications | interventions — Prednisolone; Tobramycin; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone and Tobramycin (Experimental): Prednisolone acetate 1.0% and tobramycin 0.3% ophthalmic suspension. One drop of test agent will be instilled in the inferior cul de sac of the operative eye prior to cataract extraction.
  Interventions: Drug: Prednisolone and Tobramycin
- Prednisolone (Active Comparator): Prednisolone acetate 1.0% ophthalmic suspension. One drop of test agent will be instilled in the inferior cul de sac of the operative eye prior to cataract extraction.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone and Tobramycin
  Arms: Prednisolone and Tobramycin
Drug: Prednisolone
  Other Names: Pred Forte
  Arms: Prednisolone

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of the combination test agent, prednisolone acetate 1.0% and tobramycin 0.3% ophthalmic suspension compared to PredForte (prednisolone acetate 1.0%) ophthalmic suspension. Bioequivalence will be measured by comparing aqueous humor concentrations of prednisolone acetate.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract surgery
* Avoid disallowed medications throughout study

Exclusion Criteria:

* Contraindications to the use of the test agents
* Known allergy or sensitivity to the test agents or components
* History of steroid response following topical administration of corticosteroids in the eye
* Wore contact lenses 48 hours prior to Visit 1
* An intraocular pressure that is greater than 22 mmHg or less than 5 mmHg in either eye
* Any significant illness that could be expected to interfere with study
* Used ophthalmic, topical or systemic corticosteroids or an immunomodulator for 7 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2005-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence will be measured by comparing aqueous humor concentrations of prednisolone acetate at various time points | 2 days
  Comparison of aqueous humor concentrations of prednisolone acetate at various time points

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Donald E. Beahm, MD, Great Bend, Kansas
  - Cornea Consultants/Laser Eye Consultants of Boston, Boston, Massachusetts
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - Texan Eye Care PA, Austin, Texas
  - Houston Eye Associates, Houston, Texas